CLINICAL TRIAL: NCT06753097
Title: Continuous Finger-cuff Arterial Pressure Monitoring and Intraoperative Hypotension During Non-cardiac Surgery: the Randomized DETECT II Trial
Acronym: DETECT II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Karim Kouz, MD, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-101349-BO-ff
Record Dates: First submitted 2024-12-21; First posted 2024-12-31 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Intraoperative Hypotension
Keywords: finger-cuff; blood pressure; intraoperative hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent oscillometric arterial pressure monitoring (No Intervention): In patients assigned to intermittent oscillometric arterial pressure monitoring, oscillometric arterial pressure measurements will be displayed on the patient monitor and the treating anesthesiologist will be blinded to continuous finger-cuff arterial pressure monitoring. Oscillometric arterial pressure monitoring will be performed in 2.5 minutes intervals, but clinicians are free to perform additional measurements at any time.
- Continuous finger-cuff arterial pressure monitoring (Experimental): In patients assigned to continuous finger-cuff arterial pressure monitoring, arterial pressure waveforms and measurements from the finger-cuff will be displayed on the patient monitor and treating anesthesiologists will be blinded to intermittent oscillometric arterial pressure monitoring.
  Interventions: Device: Continuous finger-cuff arterial pressure monitoring

INTERVENTIONS:
Device: Continuous finger-cuff arterial pressure monitoring — Arterial pressure will be monitored using continuous non-invasive finger-cuff arterial pressure monitoring.
  Arms: Continuous finger-cuff arterial pressure monitoring

SUMMARY:
This is a randomized trial (1) investigating whether continuous finger-cuff - compared to intermittent oscillometric - arterial pressure monitoring reduces the amount of intraoperative hypotension (specifically, from the start of induction of general anesthesia until the end of surgery) in low-to-moderate risk patients having elective non-cardiac surgery.

DETAILED DESCRIPTION:
not provided

ELIGIBILITY:
We will include three types of patients:

1. Patients scheduled for ambulatory (outpatient) elective non-cardiac surgery expected to last ≥30 minutes
2. Low-risk patients (ASA I+II) having inpatient elective non-cardiac surgery expected to last ≥60 minutes
3. Moderate-risk patients (ASA III) having inpatient elective non-cardiac surgery expected to last ≥60 minutes

We will only include patients who are 18 years or older; who will have general anesthesia; and in whom intermittent arterial pressure monitoring with upper-arm cuff oscillometry is planned.

Patients that meet one or more of the following exclusion criteria cannot participate in the trial:

* Emergency surgery
* Patients on renal replacement therapy
* Contraindications for finger-cuff monitoring (e.g., Raynaud disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Time-weighted average mean arterial pressure <65 mmHg | during the start of induction of general anesthesia until the end of surgery

SECONDARY OUTCOMES:
Time-weighted average mean arterial pressure <60 mmHg | during the start of induction of general anesthesia until the end of surgery
Time-weighted average mean arterial pressure <50 mmHg | during the start of induction of general anesthesia until the end of surgery
Time-weighted average mean arterial pressure <40 mmHg | during the start of induction of general anesthesia until the end of surgery
Absolute number of patients with at least one 1-minute episode of a mean arterial pressure <65 mmHg | during the start of induction of general anesthesia until the end of surgery
Absolute number of patients with at least one 1-minute episode of a mean arterial pressure <60 mmHg | during the start of induction of general anesthesia until the end of surgery
Absolute number of patients with at least one 1-minute episode of a mean arterial pressure <50 mmHg | during the start of induction of general anesthesia until the end of surgery
Absolute number of patients with at least one 1-minute episode of a mean arterial pressure <40 mmHg | during the start of induction of general anesthesia until the end of surgery
Cumulative duration of a mean arterial pressure <65 mmHg | during the start of induction of general anesthesia until the end of surgery
Time-weighted average mean arterial pressure >100 mmHg | during the start of induction of general anesthesia until the end of surgery
Time-weighted average mean arterial pressure >110 mmHg | during the start of induction of general anesthesia until the end of surgery
Time-weighted average mean arterial pressure >120 mmHg | during the start of induction of general anesthesia until the end of surgery
Time-weighted average mean arterial pressure >140 mmHg | during the start of induction of general anesthesia until the end of surgery

OTHER OUTCOMES:
Acute kidney injury | Up until the first postoperative day
  Acute kidney injury (binary outcome) will be defined as an increase in postoperative serum creatinine from baseline of at least 0.3 mg/dl or ≥50%.
Acute myocardial injury | Up until the first postoperative day
  Acute myocardial injury (binary outcome) will be defined based on the definition of "myocardial injury and infarction associated with non-cardiac procedures" according to the Fourth Universal Definition of Myocardial Infarction (2018)
Time-weighted average of the percentage decrease in regional cerebral oxygen saturation from the baseline | during the start of induction of general anesthesia until the end of surgery
Incidence of cerebral hypoxia | during the start of induction of general anesthesia until the end of surgery
  Cerebral hypoxia will be defined as a regional cerebral oxygen saturation (rcSO2) <50% or a decrease in rcSO2 >20% from baseline (if the baseline was ≥50%) or a decrease in rcSO2 >15% from baseline (if the baseline was <50%).
Cumulative duration of cerebral hypoxia | during the start of induction of general anesthesia until the end of surgery
  Cerebral hypoxia will be defined as a regional cerebral oxygen saturation (rcSO2) <50% or a decrease in rcSO2 >20% from baseline (if the baseline was ≥50%) or a decrease in rcSO2 >15% from baseline (if the baseline was <50%).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No